CLINICAL TRIAL: NCT06930248
Title: Efficacy of Platelet-rich Plasma in Management of Anosmia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Nasr Mohamed Ibrahim, Specialist Otorhinolaryngology department Qena General hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-24-04-02MD
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Anosmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): all patients who suffer from anosmia
  Interventions: Biological: Platelet rich plasma injection

INTERVENTIONS:
Biological: Platelet rich plasma injection — Our first step is the local anesthesia using a solution of decongestion nasal drops with 5% Emla and 10% Xylocaine spray in cotton, which is placed in the nose for 30 minutes. The 2nd step of the administration is the PRP injection in the olfactory area of the noseVia1 ml syringe with 30 G needle, PRP is injected in the olfactory area(located at superior turbinate and superior portion of lateral an medial portion of nasal cavity) approximately every 1 cm2 with the help of a nasal endoscope. The procedure is repeated 3 times with a 4 week interval with follow up patients for 6 months. A 4th time is injected after 3 months.

SUMMARY:
Olfactory dysfunction is a prevalent disorder that affects up to 20% of the general population and has significant effects on a person's quality of life as well as increased morbidity and mortality (Croy I et al., 2014;Nordin S et al

.,2008). Anosmia is the inability to perceive the odor or a lack of functioning olfaction; it may be temporary or permanent. Organic anosmia is loss of smell due to nasal obstruction caused by sinonasal diseases (as nasal polyps, tumors, postoperative) preventing odorant molecules from reaching olfactory mucosa. Functional anosmia affects up to 5% of the general population and 10% of those older than 65 . Functional anosmia is due to damage of peripheral olfactory area causing permanent loss of smell as post-traumatic, post viral infection. . 20% of individuals aged 20 to 90 years have impaired olfactory Function . The etiology of olfactory dysfunction is quite varied, including post viral posttraumatic, and idiopathic loss of smell. Unfortunately, with these etiologies, the likelihood of spontaneous recovery is generally poor with only approximately one-third of people regaining function and the duration of loss negatively correlating with recovery rate . Treatment for olfactory dysfunction is also limited. Best evidence studies recommend olfactory training and topical steroid nasal irrigations as potential therapeutics, yet both have limited efficacy . PRP is an autologous materials known to have anti-inflammatory and proregenerative properties including up regulation of growth factors including transforming growth factor, vascular endothelial growth factor, epidermal growth factor, and insulin-like growth factor. It has been used as a safe therapy effective in treating inflammation, wound healing, and peripheral neuropathies in other clinical settings. In particular, PRP has been shown to promote axon regeneration and neuroregeneration .

ELIGIBILITY:
Inclusion Criteria:

* sex:both gender.
* UPSIT score up to 10 of 40
* all patients who suffer from anosmia
* normal airway passage
* CT free of any sinonasal obstrucive lesions.

Exclusion Criteria:

* Age: below 18 years old and above 50years old.
* All patients with bilateral nasal obstruction related to chronic sinusitis, bilateral nasal polyposis,septum ,turbinate hypertrophy,tumors.
* UPSIT score more than 10 of 40.
* Traumatic causes of anosmia.
* All patients with medical history of blood diseases and diabetic and hypertensive patients.
* any medical treatment affect coagulation or bone marrow for 2 weeks prior to testing ..

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
degree of regaining olfactory function using N-butanol threshold test | Using N-butanol or 2-phenylethanol,the 2-phenylethanol has arose smell and a longer expiration date (1.5 year) while the n-butanol has an alcohol like smell and expiration date (7-8months) as it is very volatile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Croy I, Nordin S, Hummel T. Olfactory disorders and quality of life--an updated review. Chem Senses. 2014 Mar;39(3):185-94. doi: 10.1093/chemse/bjt072. Epub 2014 Jan 15. PMID 24429163
- [Background] Nordin S, Bramerson A. Complaints of olfactory disorders: epidemiology, assessment and clinical implications. Curr Opin Allergy Clin Immunol. 2008 Feb;8(1):10-5. doi: 10.1097/ACI.0b013e3282f3f473. PMID 18188011
- [Background] Landis BN, Konnerth CG, Hummel T. A study on the frequency of olfactory dysfunction. Laryngoscope. 2004 Oct;114(10):1764-9. doi: 10.1097/00005537-200410000-00017. PMID 15454769
- [Background] Murphy C, Schubert CR, Cruickshanks KJ, Klein BE, Klein R, Nondahl DM. Prevalence of olfactory impairment in older adults. JAMA. 2002 Nov 13;288(18):2307-12. doi: 10.1001/jama.288.18.2307. PMID 12425708